CLINICAL TRIAL: NCT03782350
Title: Outcome Impact of Different Tranexamic Acid Regimen in Cardiac Surgery With Cardiopulmonary Bypass (the OPTIMAL Study)
Brief Title: Outcome Impact of Different Tranexamic Acid Regimen in Cardiac Surgery With Cardiopulmonary Bypass
Acronym: OPTIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Director, the department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: the OPTIMAL study
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Homeostasis; Cardiac Surgery
Keywords: Tranexamic Acid; Antifibrinolytics; Mortality and Morbidity; Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The subject will be assigned to either high dose regimen group or low dose regimen group of tranexamic acid in a blinded fashion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care provider, investigator and outcomes assessor will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Dosage 1 (Experimental): A bolus of 30 mg/kg Tranexamic Acid for 20 min followed by a maintenance dose of 16 mg/kg/h Tranexamic Acid until the end of surgery, and a pump prime dose 2 mg/kg.
  Interventions: Drug: Tranexamic Acid Dosage 1
- Tranexamic Acid Dosage 2 (Active Comparator): A bolus of 10 mg/kg Tranexamic Acid for 20 min followed by a maintenance dose of 2 mg/kg/h Tranexamic Acid until the end of surgery, and a pump prime dose 1 mg/kg.
  Interventions: Drug: Tranexamic Acid Dosage 2

INTERVENTIONS:
Drug: Tranexamic Acid Dosage 1 — Tranexamic Acid Dosage 1
  Other Names: Cyklokapron; Transamin
  Arms: Tranexamic Acid Dosage 1
Drug: Tranexamic Acid Dosage 2 — Tranexamic Acid Dosage 2
  Other Names: Cyklokapron; Transamin
  Arms: Tranexamic Acid Dosage 2

SUMMARY:
Background and Significance A growing amount of evidence linking transfusion of allogeneic blood products with negative patient outcomes and increased cost continues to drive interest into strategies and technologies that limit patient exposure to this risk. The single largest consumer of this resource continues to be cardiac surgery, with 20% of the world wide use of allogeneic blood products accounted for by this cohort. The lysine analogs tranexamic acid (TXA) has gained wide spread use in cardiac surgery as a blood-sparing agent. Mounted evidence has proved its efficacy and safety in cardiac surgery. However, the optimal dose regimen of TXA and the impact on patients' outcomes remains debated.

Study Objectives The primary objective of the study is to analyze the primary efficacy (superiority) and primary safety (non-inferiority) of the two dose regimen of tranexamic acid.. The primary efficacy endpoint includes perioperative allogeneic transfusion rate, and the primary safety endpoint includes the 30-day rate of the composite of perioperative renal dysfunction, myocardial infarction, ischaemic stroke, seizure, deep venous thrombosis, pulmonary embolism and all-cause mortality. The secondary objectives are to demonstrate the efficacy of the two dose regimens in reducing perioperative allogeneic transfusion volume, postoperative bleeding (chest tube drainage), reoperation rate, mechanic ventilation duration, ICU stay, hospital length of stay (LOS), and total hospitalization cost.

Study Endpoints The primary endpoints include efficacy and safety. The primary efficacy endpoint includes perioperative allogeneic transfusion rate, and the primary safety endpoint includes the 30-day rate of the composite of perioperative renal dysfunction, myocardial infarction, ischaemic stroke, seizure, deep venous thrombosis, pulmonary embolism, and all-cause mortality. The key secondary endpoints of the study are defined as perioperative allogeneic transfusion volume, postoperative bleeding (chest tube drainage), reoperation rate, mechanic ventilation duration, ICU stay, hospital length of stay (LOS), and total hospitalization cost.

Study Population Adult patients aged 18-70 years undergoing elective cardiac surgery with cardiopulmonary bypass are included. Totally 3008 patients will be required for this study (1504 in each of the 2 groups).

Study Design The study is a multicenter, randomised, double-blind trial. Cardiac surgery patients with cardiopulmonary bypass will be randomised to Dosage 1 regimen group or Dosage 2 regimen group of tranexamic acid.

Study Treatment The dosage regimen is implemented with dose of loading (intravenous infusion in 20 mins), maintenance (throughout the surgery), and pump prime (added into the bypass machine). The Dosage 2 regimen contains an intravenous bolus of 10 mg/kg after anesthetic induction followed by an intravenous maintenance of 2 mg/kg/h throughout the surgery, and a pump prime dose 1 mg/kg. As for the Dosage 1 regimen, the intravenous bolus and the maintenance are 30 mg/kg and 16 mg/kg/h respectively, and a pump prime dose 2 mg/kg. Patients, surgeons and research staff interviewing patients postoperatively will be blind to treatment allocation.

Statistical Considerations The study hypothesis is that the Dosage 1 regimen of tranexamic acid is superiority to the Dosage 2 regimen in the primary efficacy endpoint, while at the same time, the Dosage 1 regimen is non-inferiority to the Dosage 2 regimen in the primary safety endpoint in cardiac surgery with cardiopulmonary bypass. The sample size calculation is mainly based on the blood transfusion rate, and 30-day rate of the composite of perioperative renal dysfunction, myocardial infarction, ischaemic stroke, seizure, deep venous thrombosis, pulmonary embolism and all-cause mortality. For the primary efficacy endpoint, a sample size estimate of 1,214 randomized subjects (607 for each group) has 90% power to detect a 12.5% reduction (61.7% vs 70.5% between Dosage 1 regimen and Dosage 2 regimen ), by means of a single-sided α = 0.025 Chi-square test. For the primary safety endpoint, a sample size estimate of 2,698 randomized subjects (1349 for each group) has 90% power to detect a noninferiority margin for the difference of 5%, by means of a single-sided α = 0.025 log rank test. In order to conduct an interim analysis, the sample size in each group is 1504(10% drop-out rate) for the adjusted significance level (from 0.025 to 0.0245 in accordance with α spending function by Lan-DeMets Method). Finally, the investigators decided to enroll 3008 study patients (1:1 ratio) for the OPTIMAL trial.

DETAILED DESCRIPTION:
A face to face visit (review in hospital, or remote video interview via smart phone and social media) is required to screen the occurrence of 30-day rate of the composite endpoints of renal dysfunction, myocardial infarction,stroke, seizure, deep venous thrombosis, pulmonary embolism and all-cause mortality, specific examinations are needed to confirm the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients aged 18~70 years.
2. Patients receiving cardiac surgery with cardiopulmonary bypass
3. Written Informed consent obtained

Exclusion Criteria:

1. Acquired chromatic disorder
2. Active intravascular coagulation
3. Previous convulsion or seizure
4. Allergy or contraindication to tranexamic acid injection or its components
5. Feeding or pregnancy women
6. Terminal illness with a life expectancy of less than 3 months
7. Patients with mental or legal disability
8. Currently enrolled in another perioperative interventional study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3079 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Perioperative allogeneic RBC transfusion rate | From the operation day to the discharge, an average of 7 days
  The overall transfusion rate of allogeneic package RBC.
Composite rate of renal dysfunction, myocardial infarction,stroke, seizure, deep venous thrombosis, pulmonary embolism and all-cause mortality | 30-day postoperatively
  A face to face visit (review in hospital, or remote video interview via smart phone and social media) is required to screen the occurrence of 30-day rate of the composite endpoints of renal dysfunction, myocardial infarction,stroke, seizure, deep venous thrombosis, pulmonary embolism and all-cause mortality, specific examinations are needed to confirm the diagnosis.

SECONDARY OUTCOMES:
Perioperative allogeneic RBC transfusion volume | From the operation day to the discharge, an average of 7 days
  The overall volume of allogeneic transfused RBC
Perioperative allogeneic non-RBC transfusion volume | From the operation day to the discharge, an average of 7 days
  The overall volume of allogeneic transfused FFP，platelet，and cryoprecipitate
Perioperative allogeneic non-RBC transfusion rate | From the operation day to the discharge, an average of 7 days
  The rate of allogeneic transfused FFP，platelet，and cryoprecipitate
Postoperative bleeding volume | From the operation day to the discharge, an average of 7 days
  The total chest tube drainage postoperatively
Reoperation rate for bleeding | From the operation day to the discharge, an average of 7 days
  Reoperation due to excessive chest tube drainage or pericardial tamponade.
The duration of mechanical ventilation | from the end of the operation and the extubation, an average of 24 hours
  The time interval between the end of the operation and the extubation
Length of stay in the intensive care unit | From the end of the operation and the discharge from the intensive care unit, an average of 48 hours
  The time interval between the end of the operation and the discharge from the intensive care unit
Length of stay in hospital | From the operation day to the discharge, an average of 7 days
  The days between the operation and the discharge from the hospital
Total hospitalization cost | In hospital, an average of 7 days
  The total cost during hospitalization

OTHER OUTCOMES:
Thrombotic test | preoperative、4~8 hours postoperative、1st postoperative day、2nd postoperative day、3rd postoperative day
  D-dimer level
Correction Dimension of Electroencephalogram | 12 hours postoperatively
  A reduced correction dimension of EEG indicates seizure
Bispectral Index | From anesthetic induction until 12 hours postoperatively, an average of 18 hours
  A range of 0~100 (85~100 awake, 65~85 sedation, 40~65 anesthesia, <40 burst suppression)
Drug concentration in plasma and cerebrospinal fluid | Fourteen timepoints from anesthetic induction until 6 hours postoperatively
  Two mililiter of blood sample will be obtained from the radial artery in 8 participants in the two groups respectively. Two mililiter of cerebrospinal fluid will be obtained in 8 participants receiving aortic surgery with subarachnoid drainage in the two groups respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences， Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalisiak A, Oosterwijk E, Minniti JG, Old LJ, Scheinberg DA. A monoclonal antibody for terminal beta-galactose. Use in analysis of glycosphingolipids. Glycoconj J. 1991 Feb;8(1):55-62. doi: 10.1007/BF00731643. PMID 1726670
- [Background] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Background] Karkouti K, Wijeysundera DN, Yau TM, Beattie WS, Abdelnaem E, McCluskey SA, Ghannam M, Yeo E, Djaiani G, Karski J. The independent association of massive blood loss with mortality in cardiac surgery. Transfusion. 2004 Oct;44(10):1453-62. doi: 10.1111/j.1537-2995.2004.04144.x. PMID 15383018
- [Background] Kurt M, Tanboga IH, Isik T, Kaya A, Ekinci M, Bilen E, Can MM, Karakas MF, Bayram E, Aksakal E, Sevimli S. Comparison of transthoracic and transesophageal 2-dimensional speckle tracking echocardiography. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):26-31. doi: 10.1053/j.jvca.2011.05.014. Epub 2011 Aug 11. PMID 21835643
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] Levi M, Cromheecke ME, de Jonge E, Prins MH, de Mol BJ, Briet E, Buller HR. Pharmacological strategies to decrease excessive blood loss in cardiac surgery: a meta-analysis of clinically relevant endpoints. Lancet. 1999 Dec 4;354(9194):1940-7. doi: 10.1016/S0140-6736(99)01264-7. PMID 10622296
- [Background] Brown JR, Birkmeyer NJ, O'Connor GT. Meta-analysis comparing the effectiveness and adverse outcomes of antifibrinolytic agents in cardiac surgery. Circulation. 2007 Jun 5;115(22):2801-13. doi: 10.1161/CIRCULATIONAHA.106.671222. Epub 2007 May 28. PMID 17533182
- [Background] Butler KD, Smith JR. Mechanisms of Forssman-induced bronchospasm and their inhibition. Br J Pharmacol. 1981 May;73(1):25-32. doi: 10.1111/j.1476-5381.1981.tb16767.x. PMID 7284697
- [Background] Schneeweiss S, Seeger JD, Landon J, Walker AM. Aprotinin during coronary-artery bypass grafting and risk of death. N Engl J Med. 2008 Feb 21;358(8):771-83. doi: 10.1056/NEJMoa0707571. PMID 18287600
- [Background] Fergusson DA, Hebert PC, Mazer CD, Fremes S, MacAdams C, Murkin JM, Teoh K, Duke PC, Arellano R, Blajchman MA, Bussieres JS, Cote D, Karski J, Martineau R, Robblee JA, Rodger M, Wells G, Clinch J, Pretorius R; BART Investigators. A comparison of aprotinin and lysine analogues in high-risk cardiac surgery. N Engl J Med. 2008 May 29;358(22):2319-31. doi: 10.1056/NEJMoa0802395. Epub 2008 May 14. PMID 18480196
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- [Background] Sander M, Spies CD, Martiny V, Rosenthal C, Wernecke KD, von Heymann C. Mortality associated with administration of high-dose tranexamic acid and aprotinin in primary open-heart procedures: a retrospective analysis. Crit Care. 2010;14(4):R148. doi: 10.1186/cc9216. Epub 2010 Aug 3. PMID 20682059
- [Background] Koster A, Borgermann J, Zittermann A, Lueth JU, Gillis-Januszewski T, Schirmer U. Moderate dosage of tranexamic acid during cardiac surgery with cardiopulmonary bypass and convulsive seizures: incidence and clinical outcome. Br J Anaesth. 2013 Jan;110(1):34-40. doi: 10.1093/bja/aes310. Epub 2012 Sep 17. PMID 22986419
- [Background] Murkin JM, Falter F, Granton J, Young B, Burt C, Chu M. High-dose tranexamic Acid is associated with nonischemic clinical seizures in cardiac surgical patients. Anesth Analg. 2010 Feb 1;110(2):350-3. doi: 10.1213/ANE.0b013e3181c92b23. Epub 2009 Dec 8. PMID 19996135
- [Background] Martin K, Knorr J, Breuer T, Gertler R, Macguill M, Lange R, Tassani P, Wiesner G. Seizures after open heart surgery: comparison of epsilon-aminocaproic acid and tranexamic acid. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):20-5. doi: 10.1053/j.jvca.2010.10.007. PMID 21272777
- [Background] Koster A, Schirmer U. Re-evaluation of the role of antifibrinolytic therapy with lysine analogs during cardiac surgery in the post aprotinin era. Curr Opin Anaesthesiol. 2011 Feb;24(1):92-7. doi: 10.1097/ACO.0b013e32833ff3eb. PMID 20881484
- [Background] Schlag MG, Hopf R, Zifko U, Redl H. Epileptic seizures following cortical application of fibrin sealants containing tranexamic acid in rats. Acta Neurochir (Wien). 2002 Jan;144(1):63-9. doi: 10.1007/s701-002-8275-z. PMID 11807648
- [Background] Horrow JC, Van Riper DF, Strong MD, Grunewald KE, Parmet JL. The dose-response relationship of tranexamic acid. Anesthesiology. 1995 Feb;82(2):383-92. doi: 10.1097/00000542-199502000-00009. PMID 7856897
- [Background] Sigaut S, Tremey B, Ouattara A, Couturier R, Taberlet C, Grassin-Delyle S, Dreyfus JF, Schlumberger S, Fischler M. Comparison of two doses of tranexamic acid in adults undergoing cardiac surgery with cardiopulmonary bypass. Anesthesiology. 2014 Mar;120(3):590-600. doi: 10.1097/ALN.0b013e3182a443e8. PMID 23903022
- [Background] Dowd NP, Karski JM, Cheng DC, Carroll JA, Lin Y, James RL, Butterworth J. Pharmacokinetics of tranexamic acid during cardiopulmonary bypass. Anesthesiology. 2002 Aug;97(2):390-9. doi: 10.1097/00000542-200208000-00016. PMID 12151929
- [Background] Grassin-Delyle S, Tremey B, Abe E, Fischler M, Alvarez JC, Devillier P, Urien S. Population pharmacokinetics of tranexamic acid in adults undergoing cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2013 Dec;111(6):916-24. doi: 10.1093/bja/aet255. Epub 2013 Jul 23. PMID 23880099
- [Background] Fiechtner BK, Nuttall GA, Johnson ME, Dong Y, Sujirattanawimol N, Oliver WC Jr, Sarpal RS, Oyen LJ, Ereth MH. Plasma tranexamic acid concentrations during cardiopulmonary bypass. Anesth Analg. 2001 May;92(5):1131-6. doi: 10.1097/00000539-200105000-00010. PMID 11323334
- [Background] Nuttall GA, Gutierrez MC, Dewey JD, Johnson ME, Oyen LJ, Hanson AC, Oliver WC Jr. A preliminary study of a new tranexamic acid dosing schedule for cardiac surgery. J Cardiothorac Vasc Anesth. 2008 Apr;22(2):230-5. doi: 10.1053/j.jvca.2007.12.016. PMID 18375325
- [Background] Du Y, Xu J, Wang G, Shi J, Yang L, Shi S, Lu H, Wang Y, Ji B, Zheng Z. Comparison of two tranexamic acid dose regimens in patients undergoing cardiac valve surgery. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1233-7. doi: 10.1053/j.jvca.2013.10.006. Epub 2014 Jan 18. PMID 24447498
- [Derived] Li Q, Lv H, Chen Y, Shen J, Shi J, Zhou C, Yan F. Development and validation of a machine learning prediction model for perioperative red blood cell transfusions in cardiac surgery. Int J Med Inform. 2024 Apr;184:105343. doi: 10.1016/j.ijmedinf.2024.105343. Epub 2024 Jan 26. PMID 38286086
- [Derived] Patel PA, Wyrobek JA, Butwick AJ, Pivalizza EG, Hare GMT, Mazer CD, Goobie SM. Update on Applications and Limitations of Perioperative Tranexamic Acid. Anesth Analg. 2022 Sep 1;135(3):460-473. doi: 10.1213/ANE.0000000000006039. Epub 2022 Aug 17. PMID 35977357
- [Derived] Shi J, Zhou C, Pan W, Sun H, Liu S, Feng W, Wang W, Cheng Z, Wang Y, Zheng Z; OPTIMAL Study Group. Effect of High- vs Low-Dose Tranexamic Acid Infusion on Need for Red Blood Cell Transfusion and Adverse Events in Patients Undergoing Cardiac Surgery: The OPTIMAL Randomized Clinical Trial. JAMA. 2022 Jul 26;328(4):336-347. doi: 10.1001/jama.2022.10725. PMID 35881121
- [Derived] Shi J, Zhou C, Liu S, Sun H, Wang Y, Yan F, Pan W, Zheng Z. Outcome impact of different tranexamic acid regimens in cardiac surgery with cardiopulmonary bypass (OPTIMAL): Rationale, design, and study protocol of a multicenter randomized controlled trial. Am Heart J. 2020 Apr;222:147-156. doi: 10.1016/j.ahj.2019.09.010. Epub 2019 Oct 21. PMID 32062173